CLINICAL TRIAL: NCT03435497
Title: Game Changers: Pilot Intervention to Empower HIV Clients as Prevention Advocates in Uganda
Brief Title: Pilot Intervention to Empower HIV Clients as Prevention Advocates in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Infectious Diseases Institute, Uganda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH111460 (NIH)
Record Dates: First submitted 2018-02-08; First posted 2018-02-19 (Actual); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-05

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game Changers Intervention (Experimental): Game Changers is an intervention that aims to empower and mobilize people living with HIV to be agents for HIV prevention and behavioral change in their social networks.
  Interventions: Behavioral: Game Changers
- Control (No Intervention): The control group will receive standard of care during the intervention assessment period. All control participants will be offered the Game Changers program once all assessments for the primary study outcomes have been completed.

INTERVENTIONS:
Behavioral: Game Changers — Game Changers is an intervention that aims to empower and mobilize PLHA to be agents for HIV prevention and behavioral change in their social networks.
  Arms: Game Changers Intervention

SUMMARY:
This randomized controlled pilot study of the "Game Changers" program will:

1. Assess the feasibility and acceptability of implementing an HIV prevention advocacy intervention with people living with HIV who are in HIV care, and who will be trained to be advocates of HIV protective behaviors within their social networks.
2. Assess preliminary intervention effects on a) protective behavior of the HIV-positive clients (condom use, partner concurrency/number of partners, engagement in HIV care, ART adherence); and b) diffusion of prevention messages across the network, as assessed by the content and extent of communication with network members about protective behaviors (condom use, partner concurrency/number of partners, HIV testing, engagement in HIV care, circumcision), HIV disclosure, and HIV stigma.
3. Explore characteristics of HIV-positive clients who more effectively engage in prevention advocacy (in terms of socio-demographics, network characteristics, and network position and type of alters receiving advocacy).

DETAILED DESCRIPTION:
People living with HIV (PLWH) have a critical role to play in HIV prevention, not only in the context of Prevention for Positives and Treatment as Prevention, but as powerful change agents for HIV protective behaviors among others. Our research suggests that as PLWH receive HIV treatment and restore their health and functioning, many are motivated to protect their loved ones and engage in prevention advocacy (i.e., to encourage friends and family to seek HIV testing and treatment, and to reduce risk behavior); however, the quality of this advocacy is hampered by challenges related to message content, style and timing of delivery, and selection of advocacy recipients. With effective advocacy training, mobilizing PLWH to be change agents within their social networks has the potential to be a "game changer" for HIV prevention, particularly in high prevalence settings such as Uganda, where virtually every family is touched by someone living with HIV. Drawing upon theoretical frameworks for network-based interventions, such as theories of social diffusion, cognitive consistency, and social influence, the proposed study will develop and pilot test "Game Changers"-- an intervention that aims to empower and mobilize PLWH to be agents for HIV prevention and behavioral change in their social networks. In Phase 1, separate focus groups of PLWH and members of their social networks (family and friends) were conducted to explore barriers to and facilitators of mobilizing clients to advocate for HIV prevention, perceptions on how advocacy could be most effective in motivating behavior change, and how to best structure the intervention and its content. In Phase 2 findings from Phase 1 and network-based intervention models were used to develop the structure and content of an intervention designed to help clients cope with stigma, manage their disease, live positively, and develop motivation and skills for HIV disclosure and prevention advocacy. In Phase 3 a pilot group intervention will be conducted in a controlled trial of 96 clients, with 48 randomly assigned to receive the intervention and 48 to the wait-list control. Assessments will be administered to all participants at baseline, 5 months later, and again 8 months after baseline, after which the control group will receive the intervention (but not the interviews). PLWH interviews and social network assessments will examine intervention effects on protective behaviors of the participant (condom use, HIV treatment adherence), and diffusion of prevention messages across the network, as assessed by the content and extent of communication with network members about protective behaviors (condom use, partner concurrency/number of partners, HIV testing, engagement in HIV care, circumcision), HIV disclosure, and HIV stigma. At the end of the intervention period a focus group with program participants will be conducted to get feedback on the intervention. To help understand how participation in the program might affect health, date of HIV diagnosis, last two CD4 counts and HIV viral loads, and prescribed HIV medications will be obtained from PLWH participant medical charts. Participants (about 15/arm) will be asked to recruit up to 3 alters each, who know the participant's serostatus, to be interviewed to assess their HIV protective behaviors (e.g., condom use) and receipt of prevention advocacy from the intervention participant.

ELIGIBILITY:
Inclusion Criteria (People living with HIV):

* 18+ years old
* In HIV care for > 1 year
* Having disclosed serostatus to at least one person

Inclusion Criteria (Social network members):

* 18+ years old
* Referred by a patient participant because they are family members, friends, or other people in patients' social network
* knows patient participant's serostatus

Exclusion Criteria:

* Individuals who meet the inclusion criteria above will be eligible to participate, and no other exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bogart, PhD, Principal Investigator — RAND
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 control was withdrawn because she was exposed to the intervention after randomization. Of the 98 remaining, 1 control did not provide any follow-up data due to moving away from the study area. 4 participants who provided first follow-up data did not provide last follow-up data (2 intervention, 2 control). Retention rate=99%
Period: Overall Study
Arm/Group | Game Changers Intervention | Control
Started | 51 | 47
Completed | 49 | 41
Not Completed | 2 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Wrong survey administered | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Game Changers Intervention | Control | Total
Number analyzed (Participants) | 51 | 47 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (10.7) | 37.1 (10.0) | 35.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 24 | 22 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 51 | 47 | 98
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 51 | 47 | 98
Engagement HIV Prevention Advocacy [Mean (Standard Deviation); unit: units on a scale] — Self-reported communication with social network members about protective behaviors: participants asked how much they discussed eight different topics (e.g., HIV testing, condom use) with people they know in the past 3 months, from 1, not at all to 5, very much
  units on a scale | 4.1 (0.9) | 3.8 (1.0) | 4.0 (1.0)
Internalized HIV Stigma [Mean (Standard Deviation); unit: units on a scale (1-5)] — Composite of 6 survey items rated on a scale of 1 (low) to 5 (high)
  units on a scale (1-5) | 1.7 (0.7) | 1.8 (0.8) | 1.8 (0.7)
Disclosure to main partner/spouse [Count of Participants; unit: Participants] | 46 | 45 | 91
HIV Treatment Adherence Percentage [Mean (Standard Deviation); unit: mean % of prescribed medication taken] — Self-reported percentage of prescribed HIV antiretroviral medications taken in the past month
  mean % of prescribed medication taken | 0.9 (0.1) | .9 (.1) | .9 (.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Engagement HIV Prevention Advocacy
Description: Self-reported communication with social network members about protective behaviors. This is a composite of 14 survey items rated on a scale of 1 (low level of communication) to 5 (high level of communication).
Time Frame: Past 3 months, measured at baseline and 5 and 8 months post-baseline
Population: 1 control participant did not provide any follow-up data due to moving away from the study area. 2 intervention and 2 control participants who provided follow-up data at 5-months post-baseline did not provide follow-up data at 8-months post-baseline. The retention rate for any follow-up data was 99%, and at last follow-up was 95%.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Game Changers Intervention | Control
Number analyzed (Participants) | 51 | 46
units on a scale
  Baseline | 4.1 (0.9) | 3.8 (1.0)
  5-Month Followup: number analyzed (Participants) | 51 | 44
  5-Month Followup | 4.2 (0.9) | 3.5 (1.1)
  8-month Followup: number analyzed (Participants) | 49 | 44
  8-month Followup | 4.0 (1.0) | 3.6 (1.0)
Statistical Analysis 1: Comparison: Game Changers Intervention vs Control; Test type: Superiority — Using an intent-to-treat approach, intervention efficacy was tested with a hierarchical linear repeated-measures regressions in which the response may have come from either follow-up, and the predictors were an indicator for study arm, the baseline value of the outcome, the follow-up time-point, and covariates. Standard errors were adjusted for clustering at the individual level (ultimate clustering methods). Covariates were socio-demographics associated with the outcome at p>.05; p = .017, Regression, Linear; Mean Difference (Net) = .4, Standard Error of Mean .2

2. Secondary Outcome: Change in Sexual Risk Behavior Among Alters
Description: Increased percentage of self-reported condom use with main partner in past 3 months
Time Frame: Measured at baseline and 5 and 8 months post-baseline
Population: We contacted 135 alters, 17 were already enrolled; 1 was withdrawn because the referring participant was exposed to the intervention. Of the remaining 117, 34 could not be reached, and 26 declined. Thus, 56 alters participated (35 referred by intervention participants, 21 referred by control). Alters were not included in the enrollment number.
Measure: Count of Participants; unit: Participants
Arm/Group | Game Changers Intervention | Control
Number analyzed (Participants) | 35 | 21
Participants
  5-Month Followup | 13 | 14
  8-month Followup | 16 | 12
Statistical Analysis 1: Comparison: Game Changers Intervention vs Control; Test type: Superiority — Using an intent-to-treat approach, intervention efficacy was tested with a hierarchical logistic repeated-measures regressions in which the response may have come from either follow-up, and the predictors were an indicator for study arm, the baseline value of the outcome, the follow-up time-point, and covariates. Standard errors were adjusted for clustering at the individual level (ultimate clustering methods). Covariates were socio-demographics associated with the outcome at p>.05; p = .05, Regression, Logistic; Mean Difference (Net) = 0.5, 95% CI 2-sided [0.2 to 1.6]

3. Secondary Outcome: Change in HIV Treatment Adherence
Description: Increased antiretroviral treatment adherence (self-reported % doses taken in past month)
Time Frame: Measured at baseline and 5 and 8 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mean % of prescribed doses taken
Arm/Group | Game Changers Intervention | Control
Number analyzed (Participants) | 50 | 46
mean % of prescribed doses taken
  Baseline | .91 (.09) | .93 (.08)
  5-Month Followup: number analyzed (Participants) | 50 | 44
  5-Month Followup | .92 (.09) | .93 (.10)
  8-month Followup: number analyzed (Participants) | 48 | 44
  8-month Followup | .95 (.06) | .93 (.12)
Statistical Analysis 1: Comparison: Game Changers Intervention vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.48, Regression, Linear; Mean Difference (Net) = 0.01, Standard Error of Mean 0.02

4. Secondary Outcome: Change in Internalized HIV Stigma
Description: Decreased rates of internalized HIV-related stigma on Internalized AIDS Stigma Scale (range=1-5, higher values = high stigma)
Time Frame: Measured at baseline and 5 and 8 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Game Changers Intervention | Control
Number analyzed (Participants) | 51 | 46
units on a scale
  Baseline | 1.7 (.7) | 1.8 (.8)
  5-Month Followup: number analyzed (Participants) | 51 | 44
  5-Month Followup | 1.6 (0.6) | 1.9 (0.7)
  8-month Followup: number analyzed (Participants) | 49 | 44
  8-month Followup | 1.4 (0.6) | 1.7 (0.8)
Statistical Analysis 1: Comparison: Game Changers Intervention vs Control; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.012, Regression, Linear; Mean Difference (Net) = -.3, Standard Error of Mean .1

5. Secondary Outcome: Number of Participants Who Have Reported Their HIV Status to Their Main Partner
Description: Increased self-reported rates of HIV status disclosure: Participants were asked if they had disclosed their HIV-serostatus to their main partner or spouse (yes/no).
Time Frame: Measured at baseline and 5 and 8 months post-baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Game Changers Intervention | Control
Number analyzed (Participants) | 31 | 30
Participants
  Baseline | 31 | 30
  5-Month Followup | 29 | 28
  8-month Followup | 31 | 27
Statistical Analysis 1: Comparison: Game Changers Intervention vs Control; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.022, Regression, Logistic; Odds Ratio (OR) = 10.0, 95% CI 2-sided [1.5 to 67.7]

ADVERSE EVENTS:
Time Frame: Approximately 1 year, 4 months (April 2018 - July 2019)
Arm/Group | Game Changers Intervention | Control
All-Cause Mortality (participants affected / at risk) | 1/51 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/47
Other Adverse Events (participants affected / at risk) | 0/51 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT03435497/Prot_SAP_001.pdf